CLINICAL TRIAL: NCT02138851
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel Trial in Subjects With Functional Constipation, to Evaluate the Improvement in Constipation of Ficus Carica
Brief Title: The Effects of a Ficus Carica in Subjects With Functional Constipation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: YGF-CON-FIG2
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Functional Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ficus Carica (Experimental): Ficus Carica 300g/day
  Interventions: Dietary Supplement: Ficus Carica (300g/day)
- Placebo (Placebo Comparator): Placebo 300g/day
  Interventions: Dietary Supplement: Placebo (300g/day)

INTERVENTIONS:
Dietary Supplement: Ficus Carica (300g/day) — Ficus Carica (300g/day), parallel design
  Arms: Ficus Carica
Dietary Supplement: Placebo (300g/day) — Placebo (300g/day), parallel design
  Arms: Placebo

SUMMARY:
The investigators performed a 8-week, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of Fig paste on functional constipation. The investigators measured colon transit time, frequency of defecation, defecation time, stool type, and abdominal discomfort.

ELIGIBILITY:
Inclusion Criteria:

* age between 19 and 39 years,
* diagnosis of functional constipation by ROME III criteria,
* Colon transit time (CTT) ≥ 36 h,
* subjects giving written informed consent

Exclusion Criteria:

* allergic or hypersensitive response to any of the ingredients in the test products,
* having previous history or current disease of digestive system, cardiovascular system, endocrine system and neurological disorder,
* diagnosis of irritable bowel syndrome by ROME III criteria, etc,.

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2013-06; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes in colon transit time | 8 weeks
  Colon transit time was measured in study baseline and visit 3(8 week). Colonic transit time was measured by the method of Metcalf et al,. Subjects ingested a once-daily series of three distinctive ColomarkTM capsules at the same time each day for three consecutive days. Each capsule contained twenty radioopaque makers of a ring shape. Subjects then received abdominal X-rays 24 after the ingestion of the ﬁnal capsule. Abdominal X-rays through a Number of markers present was confirmed. The CTT was calculated as the sum of the markers detected on X-ray.

SECONDARY OUTCOMES:
Changes in frequency of defecation | 8 week
  Frequency of defecationI was measured in study baseline and visit 3(8 week).
Changes in defecation time | 8 week
  Defecation time was measured in study baseline and visit 3(8 week).
Changes in stool type | 8 week
  Stool type was measured in study baseline and visit 3(8 week). Stool type is composed as follows: Separate hard lumps, like nuts. (score 1); Sausage-shaped but lumpy (score 2); Like a sausage or snake but with cracks on its surface (score 3); Like a sausage or snake, smooth and soft. (score 4); Soft blobs with clear-cut edges (score 5); Fluffy pieces with ragged edges, a mushy stool (score 6); Watery, no solid pieces (score 7). The average score is closer to the three-point mode means a normal stool.
Changes in abdominal discomfort | 8 week
  Abdominal discomfort was measured in study baseline and visit 3(8 week). Abdominal discomfort each question is composed as follows: Very poor (score 1); Poor (score 2); Average (score 3); Good (score 4); Very good (score 5). A higher score means severe abdominal pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea